CLINICAL TRIAL: NCT04730232
Title: An Open Label, Single-arm, Phase 2 Study of Tislelizumab Combined With Nab-Paclitaxel for Patients With High-Risk Non-Muscle-Invasive Urothelial Bladder Carcinoma Which is Not Completely Resectable
Brief Title: Tilelizumab Combined With Nab-Paclitaxel for High-Risk Non-Muscle-Invasive Urothelial Bladder Carcinoma Which is Not Completely Resectable
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Truce-02
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: High-Risk; Non-Muscle Invasive Bladder Urothelial Carcinoma
Keywords: Tislelizumab; Nab-Paclitaxel
MeSH Terms: interventions — tislelizumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab and Nab-Paclitaxel (Experimental): Tislelizumab 200mg IV on day 1 in combination with nab-paclitaxel 200mg IV on day 2 every 3 weeks for 3 or 4 cycles followed by transurethral resection biopsy.
  Interventions: Drug: Tislelizumab; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg will be administered on Day 1 of each cycle for 4 treatment cycles.
  Other Names: BGB-A317
Drug: Nab-paclitaxel — Nab-paclitaxel 200mg will be administered on Day 2 of each cycle for 4 treatment cycles.

SUMMARY:
This is a phase II study to determine the safety and efficacy of tislelizumab when given in combination with nab-paclitaxel as treatment for patients with high-risk non-muscle-invasive bladder cancer (HR NMIBC) which is not completely resectable. Patients will receive treatment with tislelizumab in combination with nab-paclitaxel every 3 weeks for 4 treatment cycles over 12 weeks followed by transurethral resection biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent;
2. Ability to comply with the protocol;
3. Age ≥ 18 years;
4. High-risk non-muscle-invasive urothelial carcinoma or high-risk non-muscle-invasive urothelial carcinoma as the main pathological component > 50%, difined as following:

   a. T1 b. High-grade Ta c.Carcinoma in situ(CIS);
5. Multi-point biopsy of bladder shows there are more than 2 section and over 3 points of pathological specimens are diagnosed as above, meanwhile, the tumor has to be diagnosed as not completely resectable by at least 2 senior urologist;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2;
7. Agreed to provide tissue examination samples (for detection of PD-L1 expression, tumor mutation load, IHC, detection of DNA and RNA, etc;)
8. Organ function level must meet the following requirements:

   * Hematological indexes: neutrophil count >= 1.5x10^9/L, platelet count >= 80x10^9/L, hemoglobin >= 6.0 g/dl (can be maintained by blood transfusion);
   * Liver function: total bilirubin <=1.5 ULN, alanine aminotransferase and aspartate aminotransferase <=2.5 ULN;
9. The subjects volunteered to join the study, signed informed consent, and had good compliance with follow-up;

Exclusion Criteria:

1. Receive live attenuated vaccine within 4 weeks before treatment or during the study period;
2. Active, known or suspected autoimmune diseases;
3. History of primary immunodeficiency;
4. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
5. Pregnant or lactating female patients;
6. Untreated acute or chronic active hepatitis B or hepatitis C infection. Under the condition of monitoring the virus copy number of patients receiving antiviral treatment, doctors can judge whether they are in line with the patients' individual conditions;
7. Prior use of immunosuppressive drugs within 4 weeks prior to the start of treatment, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroids (i.e. not more than 10 mg / day prednisolone or other corticosteroids with the same physiological dose);
8. Known or suspected allergy to tislelizumab and albumin paclitaxel;
9. Have a clear history of active tuberculosis;
10. Received PD-1 / PD-L1 / CTLA-4 antibody or other immunotherapy in the past;
11. Participating in other clinical researchers;
12. Men with reproductive capacity or women who are likely to become pregnant do not take reliable contraceptive measures;
13. Uncontrolled concurrent diseases, including but not limited to:

    * HIV infected (HIV antibody positive);
    * Severe infection in active stage or poorly controlled;
    * Evidence of serious or uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension [i.e. hypertension greater than or equal to CTCAE grade 2 after drug treatment]);
    * Patients with active bleeding or new thrombotic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-12-27 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate for tilelizumab combined with nab-paclitaxel | At the time of transurethral resection biopsy (within 9 or 12 weeks of the first dose of tislelizumab)

SECONDARY OUTCOMES:
Cystectomy-Free Survival (CFS) | up to 3 years
  defined from D1 of treatment until cystectomy.
Duration of Response (DOR) | up to 3 years
Number of adverse events and severity by grade (CTCAE) | 12 weeks of treatment plus 30 days for toxicity followup
  Safety and toxicity will be characterized according to the reported adverse event (AE) profile using NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0, as well as a patient questionnaire derived from the Patient Reported Outcomes (PRO)-CTCAE and Patient Reported Outcomes Measurement Information System (PROMIS).

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Hu, MD,PhD, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China